CLINICAL TRIAL: NCT00002517
Title: IDA VS MTZ IN INDUCTION AND INTENSIFICATION TREATMENT OF AML OR MDS IN CHILDREN, A PHASE III RANDOMIZED STUDY
Brief Title: Combination Chemotherapy in Treating Children With Newly Diagnosed Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000078212; EORTC-58921
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2002-12

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: childhood myelodysplastic syndromes; untreated childhood acute myeloid leukemia and other myeloid malignancies; childhood acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia with maturation (M2); childhood acute myelomonocytic leukemia (M4); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; childhood acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic | interventions — Cytarabine; Daunorubicin; Dexamethasone; Etoposide; Idarubicin; Mitoxantrone; Thioguanine; Radiotherapy

INTERVENTIONS:
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: dexamethasone
Drug: etoposide
Drug: idarubicin
Drug: mitoxantrone hydrochloride
Drug: thioguanine
Procedure: allogeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known which regimen of combination chemotherapy is more effective for acute myeloid leukemia or myelodysplastic syndrome.

PURPOSE: Randomized phase III trial to compare the effectiveness of different combination chemotherapy regimens in treating children who have newly diagnosed acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of idarubicin vs mitoxantrone in induction and first intensification in terms of achieving and maintaining complete remissions in children with acute myeloid leukemia or myelodysplastic syndrome.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center and disease type (de novo acute myeloid leukemia (AML) vs AML secondary to myelodysplastic syndrome (MDS) vs MDS).

* Induction: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive cytarabine (ARA-C) IV continuously on days 1 and 2 and then IV over 30 minutes every 12 hours on days 3-8, mitoxantrone IV on days 3-5, etoposide (VP-16) IV over 1 hour on days 6-8, and ARA-C intrathecally (IT) on days 1 and 8.
  * Arm II: Patients receive ARA-C and VP-16 as in arm I and idarubicin IV on days 3-5.

Patients on both arms with CNS disease at presentation receive ARA-C IT every 3 days until the CSF clears and then weekly until the first intensification. After induction, patients on both arms proceed to first intensification, regardless of response.

* First intensification: When blood counts recover and within 40 days after initiating induction, patients are randomized to 1 of 2 treatment arms.

  * Arm III: Patients receive high-dose ARA-C IV over 3 hours every 12 hours on days 1-3 (if allogeneic bone marrow transplantation (BMT) is planned) or days 1-4 (if allogeneic BMT is not planned) and mitoxantrone IV on days 7-9.
  * Arm IV: Patients receive high-dose ARA-C as in arm III and idarubicin IV on days 7-9.
* Patients who achieve complete remission (CR) after first intensification and have an HLA-identical, chronic myelomonocytic leukemia-nonreactive, sibling donor undergo allogeneic BMT. Patients who achieve CR after intensification and have no suitable donor receive intensive chemotherapy as defined below. All patients with chloroma at presentation undergo local radiotherapy beginning after final intensification.
* Second intensification: When blood counts recover, patients receive daunorubicin IV continuously, ARA-C IV continuously, VP-16 IV continuously, oral thioguanine, and oral dexamethasone on days 1-4 and 11-14 and ARA-C IT on days 1, 4, 11, and 14.
* Third intensification: When blood counts recover, patients receive high-dose ARA-C IV over 3 hours every 12 hours on days 1-3 and VP-16 IV over 1 hour on days 2-5. When blood counts recover, autologous bone marrow is harvested in the event of subsequent relapse.
* Maintenance: When blood counts recover, patients receive oral thioguanine daily and ARA-C subcutaneously 4 days a month for 1 year.

PROJECTED ACCRUAL: A total of 310 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute myeloid leukemia (AML) based on the cytological, cytochemical, and immunological criteria of the FAB classification

  * Must meet 1 of the following criteria:

    * More than 30% blasts in marrow (calculation based on the total number of nucleated cells except lymphocytes and plasmocytes)
    * Presence of granulocytic sarcoma (chloroma)
  * Disease must be associated with at least 1 of the following:

    * More than 3% myeloperoxidase- or Sudan black-positive blasts
    * More than 3% platelet peroxidase-positive blasts
    * More than 20% esterase-positive blasts
    * Immunological markers compatible with a myeloid differentiation, including 1 of the following criteria:

      * Blasts positive for myeloid-associated antigen and negative for B- or T-lymphocyte antigens
      * Blasts positive for at least 2 myeloid antigens (except CD3 and CD8)
    * A cytogenetic abnormality associated with AML OR
* Newly diagnosed myelodysplastic syndrome (MDS) based on the cytological and cytochemical criteria of the FAB classification

  * Eligible subtypes:

    * Refractory anemia with excess blasts (RAEB)
    * RAEB in transformation
    * Chronic myelomonocytic leukemia
* No promyelocytic leukemia (M3 or M3v) treated with tretinoin (protocol EORTC-06915)
* No AML secondary to hematologic or malignant disease other than MDS
* Registration must occur within 48 hours of diagnosis

PATIENT CHARACTERISTICS:

Age:

* Under 15

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* No uncontrolled bleeding disorder

Hepatic:

* Not specified

Renal:

* No renal failure

Cardiovascular:

* No congenital heart disease

Other:

* No encephalopathy
* No genetic disorders
* No uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior antileukemic therapy

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1993-03; Primary Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Behar, MD, Study Chair — Hopital Americain
Locations (23):
- Belgium (7):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Hopital Universitaire Des Enfants Reine Fabiola, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - U.Z. Gasthuisberg, Leuven
  - Centre Hospitalier Regional de la Citadelle, Liège
  - Clinique de l'Esperance, Montegnée
- France (15):
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - CHR de Besancon - Hopital Saint-Jacques, Besançon
  - CHU de Caen, Caen
  - CHR de Grenoble - La Tronche, Grenoble
  - Centre Hospitalier Regional de Lille, Lille
  - Hopital Debrousse, Lyon
  - Hopital Arnaud de Villeneuve, Montpellier
  - CHR Hotel Dieu, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital Robert Debre, Paris
  - Institut Curie - Section Medicale, Paris
  - Hopital Jean Bernard, Poitiers
  - Hopital Americain, Reims
  - Hopital Universitaire Hautepierre, Strasbourg
  - Hopital des Enfants (Purpan Enfants), Toulouse
- Hospital Escolar San Joao, Porto, Portugal

REFERENCES:
- [Result] Brunet AS, Ploton C, Galambrun C, Pondarre C, Pages MP, Bleyzac N, Freydiere AM, Barbe G, Bertrand Y. Low incidence of sepsis due to viridans streptococci in a ten-year retrospective study of pediatric acute myeloid leukemia. Pediatr Blood Cancer. 2006 Nov;47(6):765-72. doi: 10.1002/pbc.20706. PMID 16333838
- [Result] Entz-Werle N, Suciu S, van der Werff ten Bosch J, Vilmer E, Bertrand Y, Benoit Y, Margueritte G, Plouvier E, Boutard P, Vandecruys E, Ferster A, Lutz P, Uyttebroeck A, Hoyoux C, Thyss A, Rialland X, Norton L, Pages MP, Philippe N, Otten J, Behar C; EORTC Children Leukemia Group. Results of 58872 and 58921 trials in acute myeloblastic leukemia and relative value of chemotherapy vs allogeneic bone marrow transplantation in first complete remission: the EORTC Children Leukemia Group report. Leukemia. 2005 Dec;19(12):2072-81. doi: 10.1038/sj.leu.2403932. PMID 16136166